CLINICAL TRIAL: NCT02631642
Title: A Phase I,Randomized,Double Blinded,Placebo-controlled,Dose-escalating Study of the Safety,Tolerability and Pharmacokinetics of HMPL-689 in Healthy Volunteers
Brief Title: A Study of HMPL-689 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2015-689-00AU2
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HMPL-689 (Experimental): Subjects will receive a single dose of HMPL-689 or matching placebo on Day 1. The planned dose levels in ascending order are: 1, 2.5, 5, 10, 20, 25 and 30 mg (7 dose cohorts with 8 subjects in each cohort). Within each cohort, randomization ratio of 3:1 is followed to dose 6 subjects with HMPL-689 and 2 subjects with placebo.
  Interventions: Drug: HMPL-689
- HMPL-689 placebo (Placebo Comparator): Subjects will receive a single dose of HMPL-689 or matching placebo on Day 1. The planned dose levels in ascending order are: 1, 2.5, 5, 10, 20, 25 and 30 mg (7 dose cohorts with 8 subjects in each cohort). Within each cohort, randomization ratio of 3:1 is followed to dose 6 subjects with HMPL-689 and 2 subjects with placebo.
  Interventions: Drug: HMPL-689 placebo

INTERVENTIONS:
Drug: HMPL-689 — selective PI3Kδ inhibitor
  Other Names: Huchison Medipharma
  Arms: HMPL-689
Drug: HMPL-689 placebo — placebo of HMPL-689
  Other Names: Huchison Medipharma
  Arms: HMPL-689 placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a single dose of HMPL-689 in healthy volunteers To determine the pharmacokinetic profile of single oral doses of HMPL-689 in healthy volunteers

DETAILED DESCRIPTION:
Subjects will receive a single dose of HMPL-689 or matching placebo during Day 1. The planned dose levels are: 1, 2.5, 5, 10, 20, 25 and 30 mg (about 7 cohorts of 8 subjects). In each dose cohort, 8 subjects will be randomized to receive HMPL-689 (6 subjects) or placebo (2 subjects) under fed condition with a standard meal.

For the first dose Cohort (1 mg), a sentinel group of 2 subjects (1 HMPL-689 and 1 placebo) will be dosed 24 hours prior to the planned dosing of the remaining six subjects. The decision of dose escalation or study termination will be made jointly by the principal investigator and the sponsor based on the clinical data (safety, tolerability, available PK data and clinical laboratory values). Any dose level may be repeated, reduced or split into 2 doses if deemed appropriate by the Principal Investigator and Sponsor's medical Expert.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be obtained in writing for all subjects before enrollment into the study
2. Healthy male subjects aged 18 to 45 years inclusive at the time of screening
3. Body mass index ≥19.0 and ≤ 30.0 kg/m2
4. Willing to comply with the contraceptive requirements of the study and must not donate sperm during the study or for 3 months afterwards. Subjects must agree to use a condom or to abstain from sexual intercourse throughout the trial and for 30 days afterwards

Exclusion Criteria:

1. Family history of premature Coronary Heart Disease
2. History of immunosuppression or opportunistic infections or receipt of a live virus vaccination within the 3 months prior to screening
3. Clinically significant abnormalities as determined by medical history physical examination, or laboratory test, especially for liver and renal function
4. Clinically significant findings in ECG, blood pressure and heart rate, as determined by the Clinical Investigator
5. Subjects at risk for tuberculosis (TB), which is defined as:

   1. Current clinical or laboratory evidence of active TB
   2. History of TB
   3. A positive QuantiFERON® test at screening or within 6 months prior to Day 1
6. Any medical condition requiring regular use of medication
7. Exposure to prescription medications within 30 days prior to Day 1
8. Exposure to any other medication, including over-the-counter medications, herbal remedies and vitamins 14 days prior to first dose (except for paracetamol)
9. Participation in another clinical trial with any investigational drug within 30 days of Day 1
10. Treatment in the previous 3 months with any drug known to have a well-defined potential for toxicity to a major organ
11. Current smoker of more than 10 cigarettes or equivalent/ day prior to commencing the study and unable to completely stop smoking during the study
12. Symptoms of a clinically significant illness in the 3 months before the study
13. Presence or sequelae of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
14. Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease, hemorrhoids or anal diseases with regular or recent presence of blood in feces
15. History of significant allergic disease (e.g. allergic to medications) and acute phase of allergic rhinitis in the previous 2 weeks before randomization/ enrollment or any food allergy
16. Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV)
17. Current evidence of drug abuse or history of drug abuse within one year before randomization/ enrollment
18. Mental condition rendering the subject incapable to understand the nature, scope, and possible consequences of the study
19. Unlikely to comply with the clinical study protocol; e.g. uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
20. Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
dose limited toxicities evaluated with NCI CTCAE v4.03 | within 28 days after the first dose
  Incidence of dose limited toxicities and associated dose of HMPL-689

SECONDARY OUTCOMES:
maximum plasma concentration calculated with Blood samples | within 29 days after the first dose
  Blood samples will be taken to measure the levels of study drug
time to reach maximum concentration calculated with Blood samples | within 29 days after the first dose
  Blood samples will be taken to measure the levels of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No